CLINICAL TRIAL: NCT04184830
Title: A Pilot Study of Improving Cognition in Schizophrenia Using Direct Current Stimulation
Brief Title: Improving Cognition in Schizophrenia Using Non-invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/LO/0248
Record Dates: First submitted 2019-11-25; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS arm (Experimental): Active stimulation:
  Direct current will be transferred using a pair of saline-soaked surface sponge electrodes (5x7). For anodal stimulation of the left DLPFC the anode will be placed over the site of F3, according to the 10-20 international system for electroencephalogram electrode placement. The cathode will be placed over the right supraorbital area. A constant current of 2mA will be applied for 30 minutes, which will result in current density of 0.08 mA/cm².In order to avoid side effects, as a result of electrical transient (e.g. tingling and burning sensation), the current will be ramped for 10 seconds at the beginning and end of stimulation (Nitsche et al., 2008).
  Interventions: Device: non-invasive brain stimulation
- tDCS sham (Sham Comparator): Sham stimulation:
  During the sham stimulation a pair of saline-soaked surface sponge electrodes (5x7) will be places on the scalp For sham stimulation of the left DLPFC the anode will be placed over the site of F3, according to the 10-20 international system for electroencephalogram electrode placement. The cathode will be placed over the right supraorbital area. A constant current of 2mA will be applied for 30 seconds.In order to avoid side effects, as a result of electrical transient (e.g. tingling and burning sensation), the current will be ramped for 10 seconds at the beginning and end of stimulation (Nitsche et al., 2008).
  Interventions: Device: non-invasive brain stimulation

INTERVENTIONS:
Device: non-invasive brain stimulation

SUMMARY:
This is a double-blind sham-controlled study to evaluate the effects of the combination of non-invasive brain stimulation, i.e. transcranial direct current stimulation (tDCS), with brief cognitive training (CT) on cognition in patients with schizophrenia. All participants will practice the same cognitive training tasks and will be randomised to either real tDCS or sham stimulation. Patients with schizophrenia will undergo the study interventions while maintaining their standard treatment with antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Treatment with stable doses of antipsychotic medications. For the purpose of this study stability is defined as a not more than 50% change in the dose of their antipsychotic medication 3 months preceding the screening visit.
* Age between 18 and 55 years
* Written and witnessed informed consent
* Participants must read and write in English at a level sufficient to understand and complete study-related procedures

Exclusion Criteria:

DSM-IV diagnosis of alcohol or drug dependence in the 6 months, current treatment with benzodiazepines or hypnotics

* Current or past skin disease
* History of a neurological disorder or a systemic illness with known neurological complications; including epilepsy
* History of seizures
* Head injury, accompanied with loss of consciousness or/and required hospitalization
* Unwillingness or inability to follow or comply with the procedures outlined in the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Does the combination of tDCS with brief working memory training will enhance the learning capacity of the research participants compared to sham stimulation, and whether the learning rates will be retained in the longer-term | 56 days
  The change in learning on a working memory training tasks will be analyzed using a full maximum likelihood-random effect multilevel models (MLREM). The MLREM will include the working memory outcome measure during the tDCS, next day retention at the session following tDCS administration and longer-term retention; controlled for baseline performance with fixed categorical effects for group (real tDCS vs sham stimulation) and time (0-4); an interaction of time and group.
Does the combination of tDCS with brief stochastic learning training will enhance the learning capacity of the research participants compared to sham stimulation, and whether the learning rates will be retained in the longer-term | 56 days
  The change in learning on a stochastic training tasks will be analyzed using a full maximum likelihood-random effect multilevel models (MLREM). The MLREM will include the stochastic learning task outcome measure during the tDCS, next day retention at the session following tDCS administration, and longer-term retention; controlled for baseline performance with fixed categorical effects for group (tDCS vs sham stimulation) and time (0-4); an interaction of time (0-4) and group.
Does the combination of tDCS with brief implicit learning training will enhance the learning capacity of the research participants compared to sham stimulation, and whether the learning rates will be retained in the longer-term | 56 days
  The change in learning on an implicit training tasks performance will be analyzed using a full maximum likelihood-random effect multilevel models (MLREM). The MLREM will include the task outcome measure during the tDCS administration, next day retention at the session following tDCS administration, and longer-term retention; controlled for baseline performance with fixed categorical effects for group (real tDCS vs sham stimulation) and time (0-3); an interaction of time (0-3) and group. The MLREM model will exclude the second acute tDCS session, as the task design was optimized fMRI.
The change in neuronal activity during a working memory task in response to real tDCS vs sham stimulation. | 1 day
  A comparison of neural blood oxygen level-dependent (BOLD) response during a working memory task in the real tDCS vs sham stimulation.
The change in neuronal activity during a stochastic learning task in response to real tDCS vs sham stimulation. | 1 day
  A comparison of neural blood oxygen level-dependent (BOLD) response during a stochastic learning task in the real tDCS vs sham stimulation.
The change in neuronal activity during an implicit learning task in response to real tDCS vs sham stimulation. | 1 day
  A comparison of neural blood oxygen level-dependent (BOLD) response during an implicit learning memory task in the real tDCS vs sham stimulation.
The change in neuronal activity during an executive functioning task response to real tDCS vs sham stimulation. | 1 day
  A comparison of neural blood oxygen level-dependent (BOLD) response during an executive function task in the real tDCS vs sham stimulation.

SECONDARY OUTCOMES:
The secondary outcome measure is going to be the generalization of learning to non-trained task. | 3 years
  The secondary outcome measure is the generalization of learning to non-trained task, indexed by the CogState neuropsychological battery. We will test if the effects of cognitive training and real tDCS would generalize onto significant performance improvements on related cognitive domains of executive function, and attention and vigilance as measured by the CogState neuropsychological assessment battery. The between group (1-realtDCS/ 0-sham stimulation) differences on these tasks will be tested using regressions, controlled for baseline performance.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orlov ND, Muqtadir SA, Oroojeni H, Averbeck B, Rothwell J, Shergill SS. Stimulating learning: A functional MRI and behavioral investigation of the effects of transcranial direct current stimulation on stochastic learning in schizophrenia. Psychiatry Res. 2022 Nov;317:114908. doi: 10.1016/j.psychres.2022.114908. Epub 2022 Oct 14. PMID 37732853